CLINICAL TRIAL: NCT03333382
Title: Plastic vs. Fully Covered Self Expanding Stents (FCSEMS) for Treatment of Anastomotic Bile Leaks Following Orthotopic Liver Transplant (OLT): a Randomized Controlled Trial
Brief Title: Plastic vs. Fully Covered Self Expanding Stents (FCSEMS) for Treatment of Anastomotic Bile Leaks
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Post transplant leaks are now less frequent at VUMC and we struggled to enroll.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Patrick Yachimski, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 171573
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Results first posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Bile Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Plastic Biliary Stent (Active Comparator): Subjects with anastomotic bile leaks following orthotopic liver transplant (OLT) will have a temporary plastic biliary stent placed across the site of the leak during retrograde cholangiopancreatography (ERCP).
  Interventions: Device: Plastic biliary stent
- FCSEMS (Active Comparator): Subjects with anastomotic bile leaks following orthotopic liver transplant (OLT) will have a temporary fully covered self-expanding metal stent (FCSEMS) placed across the site of the leak during retrograde cholangiopancreatography (ERCP).
  Interventions: Device: FCSEMS

INTERVENTIONS:
Device: Plastic biliary stent — Plastic biliary stent which functions largely as a wick to siphon bile flow from the site of anastomotic leak.
  Arms: Plastic Biliary Stent
Device: FCSEMS — FCSEMS has a relatively larger expansile diameter and membrane coating to provide an actual seal at site of anastomotic leak.
  Arms: FCSEMS

SUMMARY:
Standard endoscopic management for anastomotic bile leaks following OLT has been endoscopic retrograde cholangiopancreatography (ERCP) with placement of a temporary plastic biliary endoprosthesis (stent) across the site of anastomotic leak. While this intervention carries a high rate of technical success, clinical success is not universal. An alternative to placement of a plastic biliary stent is placement of a fully covered self-expanding metal stent (FCSEMS). Whereas a plastic stent functions largely as a wick to siphon bile flow, the theoretical advantage of a FCSEMS is that the relatively larger expansile diameter and membrane coating provide an actual and effective seal at the site of leak. FCSEMS have been used successfully for salvage therapy of anastomotic bile leaks in the post-OLT population with no serious stent related adverse events and no cases of unsuccessful FCSEMS removal in this population.

The objective of this study is to prospectively randomize patients found to have anastomotic bile leaks following OLT to placement of either a plastic biliary stent or a FCSEMS at initial ERCP intervention.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing ERCP for suspected anastomotic bile leak within 60 days following OLT with standard biliary reconstruction
* cognitively impaired population with a surrogate who has legal power of attorney

Exclusion Criteria:

* patients who have undergone OLT with hepaticojejunostomy
* patients who have undergone percutaneous transhepatic cholangiogram with percutaneous biliary intervention following OLT and prior to ERCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2020-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yachimski, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the patient population at the Vanderbilt Digestive Disease Center. 1 participant signed consent 1/30/18 and screen failed. 1 participant enrolled and randomized 8/21/18 and was lost to follow-up. No other participants enrolled. Study remained open in anticipation of enrolling more participants. Enrollment struggled because post transplant leaks have become less frequent at VUMC. In September 2020, the decision was made to close the study (low enrollment).
Pre-assignment Details: Only 1 participant was randomized. However, they were lost to follow-up. No participants completed the study.
Period: Overall Study
Arm/Group | Plastic Biliary Stent | FCSEMS
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 participant was randomized in the study. This participant was randomized to the Plastic Biliary Stent arm. No participants were randomized to the FCSEMS arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Plastic Biliary Stent | FCSEMS | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (0) |  | 62 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Cholangiographic Resolution of Bile Leak at Follow-up ECRP
Description: Adjudication of the primary study endpoint will be determined by the presence/absence of persistent anastomotic bile leak at first follow-up endoscopic retrograde cholangiopancreatography (ERCP) after initial stent placement, whether performed at 6 weeks or sooner.
Time Frame: up to 6 weeks
Population: Participant enrolled to Plastic Biliary Stent arm was lost to follow-up. No participants were randomized to the FCSEMS arm.
Arm/Group | Plastic Biliary Stent | FCSEMS
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Need for Repeat Endoscopic Intervention (ERCP) Within Initial 8 Weeks Following Placement of a Plastic Stent or FCSEMS
Description: Analysis for need of repeat endoscopic intervention (ERCP) within initial 8 weeks following placement of a plastic stent or FCSEMS will be completed.
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | Plastic Biliary Stent | FCSEMS
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Need for Percutaneous Drainage of Biloma or Intraabdominal Fluid Collection Following Placement of a Plastic Stent or FCSEMS
Description: Participants will be analyzed regarding need for percutaneous drainage of biloma or intraabdominal fluid collection following placement of a plastic stent or FCSEMS.
Time Frame: 90 days
Population: as for outcome 1
Arm/Group | Plastic Biliary Stent | FCSEMS
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Need for Surgical Biliary Reconstruction for Refractory Anastomotic Bile Leak
Description: Participants will be analyzed for need of surgical biliary reconstruction for refractory anastomotic bile leak
Time Frame: 90 days
Population: as for outcome 1
Arm/Group | Plastic Biliary Stent | FCSEMS
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Need for Repeat OLT
Description: Analysis for of need for orthotopic liver transplant (OLT) will be completed.
Time Frame: 90 days
Population: as for outcome 1
Arm/Group | Plastic Biliary Stent | FCSEMS
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Death at 90 Days
Description: Participants will be followed and chart review will be completed to see if death occurred within 90 days.
Time Frame: 90 days
Population: as for outcome 1
Arm/Group | Plastic Biliary Stent | FCSEMS
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Rate of Post-ERCP Pancreatitis (PEP) Following Placement of a Plastic Stent vs FCSEMS
Description: Analysis will be performed to determine rate of post-ERCP pancreatitis (PEP) following placement of a plastic stent vs FCSEMS.
Time Frame: 90 days
Population: as for outcome 1
Arm/Group | Plastic Biliary Stent | FCSEMS
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Rate of Stent Migration Following Placement of a Plastic Stent vs FCSEMS
Description: Analysis will be performed to determine the rate of stent migration following placement of a plastic stent vs FCSEMS.
Time Frame: 90 days
Population: as for outcome 1
Arm/Group | Plastic Biliary Stent | FCSEMS
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Rate of Anastomotic Biliary Stricture at Follow-up ERCP 8 Weeks Following Placement of a Plastic Stent or FCSEMS
Description: Rate of anastomotic biliary stricture at follow-up ERCP 8 weeks following placement of a plastic stent or FCSEMS will be analyzed during the course of the study.
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | Plastic Biliary Stent | FCSEMS
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Need for Repeat ERCP for Management of Anastomotic Biliary Stricture Within 90 Days Following Leak Resolution
Description: Participants will be analyzed for need of repeat ERCP for management of anastomotic biliary stricture within 90 days following leak resolution.
Time Frame: 90 days
Population: as for outcome 1
Arm/Group | Plastic Biliary Stent | FCSEMS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Definition of adverse event and/or serious adverse event did not differ from the clinicaltrials.gov definitions.
Arm/Group | Plastic Biliary Stent | FCSEMS
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
One participant screen failed before being randomized to either arm of the study. A second participant was enrolled in August 21, 2018 and was lost to follow-up. No other participants were enrolled. The study remained open in anticipation of enrolling more participants. Post transplant leaks have become less frequent at VUMC, and we struggled to enroll. In September 2020, the decision was made to close the study due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03333382/Prot_SAP_000.pdf